CLINICAL TRIAL: NCT03896269
Title: Phase 1 Dose Escalation Study of CPX-351 for Patients With Int-2 or High Risk IPSS Myelodysplastic Syndromes and Chronic Myelomonocytic Leukemia After Failure to Hypomethylating Agents
Brief Title: CPX-351 in Treating Patients With Relapsed or Refractory High Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0911; NCI-2019-01558 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0911 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Blasts 10-19 Percent of Bone Marrow Nucleated Cells; Blasts More Than 5 Percent of Bone Marrow Nucleated Cells; High Risk Chronic Myelomonocytic Leukemia; Recurrent Chronic Myelomonocytic Leukemia; Recurrent High Risk Myelodysplastic Syndrome; Refractory Chronic Myelomonocytic Leukemia; Refractory High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic | interventions — CPX-351; Injections; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (liposome-encapsulated daunorubicin-cytarabine) (Experimental): INDUCTION THERAPY: Patients receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. After 2-5 weeks, patients who do not achieve a CR/CRi/CRp, have acceptable or no toxicity, and have stable disease and no disease progression may receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION THERAPY: Patients who achieve at least a HI response, receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After 5-8 weeks, patients who do not show clinically significant disease progression or unacceptable toxicity may receive liposome-encapsulated daunorubicin-cytarabine for up to 12 additional cycles.
  Interventions: Drug: Liposome-encapsulated Daunorubicin-Cytarabine

INTERVENTIONS:
Drug: Liposome-encapsulated Daunorubicin-Cytarabine — Given IV
  Other Names: CPX-351; Cytarabine-Daunorubicin Liposome for Injection; Liposomal AraC-Daunorubicin CPX-351; Liposomal Cytarabine-Daunorubicin; Liposome-encapsulated Combination of Daunorubicin and Cytarabine; Vyxeos

SUMMARY:
This phase I trial studies best dose and side effects of liposome-encapsulated daunorubicin-cytarabine (CPX-351) and how well it works in treating patients with high risk myelodysplastic syndrome or chronic myelomonocytic leukemia that has come back or has not responded to treatment. Drugs used in chemotherapy, such as liposome-encapsulated daunorubicin-cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and tolerability of CPX-351 in patients with intermediate-2 or high-risk myelodysplastic syndrome (MDS). (Dose Escalation Stage) II. To determine the maximum tolerated dose (MTD) of intravenous CPX-351 in patients with intermediate-2 or high-risk MDS. (Dose Escalation Stage) III. To further characterize the safety and tolerability of CPX-351 in patients with intermediate-2 and high-risk MDS. (Dose-Expansion Stage) IV. To evaluate preliminary efficacy of CPX-351 in patients with intermediate-2 or high-risk MDS. (Dose-Expansion Stage)

SECONDARY OBJECTIVES:

I. To assess overall response (OR) rate. II. To assess overall survival. III. To assess duration of response. IV. To assess relapse-free survival. V. To assess safety profile.

OUTLINE: This is a dose-escalation study.

INDUCTION THERAPY: Patients receive liposome-encapsulated daunorubicin-cytarabine intravenously (IV) over 90 minutes on days 1, 3, and 5 in the absence of disease progression or unacceptable toxicity. After 2-5 weeks, patients who do not achieve a complete response (CR)/CR with incomplete bone marrow recovery (CRi)/CR with incomplete platelet recovery (CRp), have acceptable or no toxicity, and have stable disease and no disease progression may receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION THERAPY: Patients who achieve at least a hematological improvement (HI) response, receive liposome-encapsulated daunorubicin-cytarabine IV over 90 minutes on days 1 and 3. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After 5-8 weeks, patients who do not show clinically significant disease progression or unacceptable toxicity may receive liposome-encapsulated daunorubicin-cytarabine for up to 12 additional cycles.

After completion of study treatment, patients are followed up at 30 days and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MDS or chronic myelomonocytic leukemia (CMML) according to World Health Organization (WHO)
* Patients are either not eligible for or choose not to proceed with a stem cell transplant at the time of enrollment
* MDS and CMML classified by International Prognostic Scoring System (IPSS) as intermediate-2/high risk with excess blasts > 5%, or with 10-19% bone marrow blasts
* No response following at least 4 cycles of therapy or relapse after initial CR, partial response (PR), or HI or progression after any number of cycles of either azacitidine, decitabine, guadecitabine or ASTX727 (oral decitabine) as single agents or in combination with other investigational agents
* Patient (or patient's legally authorized representative) must have signed an informed consent document indicating that the patient understands the purpose of and procedures required for the study and is willing to participate in the study
* Total bilirubin < 3 mg/dL (will allow less than 5 x upper limit of normal [ULN] if Gilbert's at investigator's discretion)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) =< 3 x ULN
* Serum creatinine clearance > 30 mL/min and no end/stage renal disease
* Hydroxyurea for control of leukocytosis or use of hematopoietic growth factors (eg, granulocyte-colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], procrit, aranesp, thrombopoietins) is allowed at any time prior to or during study if considered to be in the best interest of the patient

Exclusion Criteria:

* New York Heart Association (NYHA) class III or IV congestive heart failure or left ventricular ejection fraction (LVEF) < 50 by echocardiogram or multigated acquisition (MUGA) scan
* History of myocardial infarction within the last 6 months or unstable/uncontrolled angina pectoris or history of severe and/or uncontrolled ventricular arrhythmias
* Uncontrolled infection not adequately responding to appropriate antibiotics
* Female patients who are pregnant or lactating
* Patients with reproductive potential who are unwilling to following contraception requirements (including condom use for males with sexual partners, and for females: prescription oral contraceptives [birth control pills], contraceptive injections, intrauterine devices [IUD], double-barrier method [spermicidal jelly or foam with condoms or diaphragm], contraceptive patch, or surgical sterilization) throughout the study
* Female patients with reproductive potential who have a positive urine or blood beta-human chorionic gonadotropin (beta HCG) pregnancy test at screening
* Patients receiving any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy (within 14 days of initiating study treatment)
* Prior cumulative anthracycline exposure of > 550 mg/m^2 daunorubicin or equivalent, or > 400 mg/m^2 in patients who received radiation therapy to the mediastinum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2019-05-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (dose-escalation stage) | Up to 30 days
  Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median, and range. Toxicity type, severity, and attribution will be summarized for each patient using frequency tables.
Maximum-tolerated dose (MTD) of liposome-encapsulated daunorubicin-cytarabine (dose-escalation stage) | Up to 28 days
  Defined as the highest dose level in which a dose-limiting toxicity (DLT) occurs within at most 1 out of 6 patients treated. DLTs are defined as any related non-hematological Common Terminology Criteria for Adverse Events grade >= 3 adverse events that prevent further administration of the agent at that same dose level.
Incidence of adverse events (dose-expansion stage) | Up to 30 days
  Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median, and range. Toxicity type, severity, and attribution will be summarized for each patient using frequency tables.
Objective response rate (ORR) (dose-expansion stage) | Up to 1.5 years
  Defined as complete response (CR), partial response, CR with incomplete bone marrow recovery, marrow CR or hematological improvement. Will be estimated along with 95% confidence intervals treated at the MTD (i.e., including those treated at the MTD during dose escalation and dose expansion phases). The association between ORR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

SECONDARY OUTCOMES:
Overall response rate | Up to 1.5 years
Overall survival | Up to 1.5 years
  The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Duration of response | Up to 1.5 years
  Will be summarized using descriptive statistics such as mean, standard deviation, median and range.
Relapse-free survival | Up to 1.5 years
  The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Incidence of adverse events | Up to 1.5 years
  Safety data of the patients will be summarized using descriptive statistics such as mean, standard deviation, median, and range. Toxicity type, severity, and attribution will be summarized for each patient using frequency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo M Bravo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Montalban-Bravo G, Jabbour E, Borthakur G, Kadia T, Ravandi F, Chien K, Pemmaraju N, Hammond D, Dong XQ, Huang X, Schneider H, John R, Kanagal-Shamana R, Loghavi S, Kantarjian H, Garcia-Manero G. Phase 1/2 study of CPX-351 for patients with Int-2 or high risk International Prognostic Scoring System myelodysplastic syndromes and chronic myelomonocytic leukaemia after failure to hypomethylating agents. Br J Haematol. 2024 Mar;204(3):898-909. doi: 10.1111/bjh.19193. Epub 2023 Nov 10. PMID 37946611
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/69/NCT03896269/ICF_000.pdf